CLINICAL TRIAL: NCT04464811
Title: Furosemide Stress Test for the Prediction of Acute Kidney Injury Severity in Acute Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kajohnsak Noppakun, Assistant Professor of Medicine, Chiang Mai University
Other Study IDs: MED-2563-07080 (1)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure; Acute Kidney Injury
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure with diuretic resistance: This group includes acute heart failure patients who has diuretic resistance from furosemide stress test. Furosemide stress test will be performed by administration of intravenous furosemide 1 mg/kg in patients who do not receive oral furosemide before and 1.5 mg/kg patients who have received oral furosemide before. Diuretic resistance was defined as urine output <250 hr at 2 hours after furosemide administration.
  Interventions: Diagnostic Test: Furosemide stress test
- Heart failure without diuretic resistance: This group includes acute heart failure patients who do not have diuretic resistance from furosemide stress test. Furosemide stress test will be performed by administration of intravenous furosemide 1 mg/kg in patients who do not receive oral furosemide before and 1.5 mg/kg patients who have never received oral furosemide before. Patients will be defined not to have diuretic resistance if their urine output ≥250 hr at 2 hours after furosemide administration.
  Interventions: Diagnostic Test: Furosemide stress test

INTERVENTIONS:
Diagnostic Test: Furosemide stress test — Furosemide stress test is performed by administration of intravenous furosemide 1 mg/kg in patients who do not receive oral furosemide before and 1.5 mg/kg patients who have never received oral furosemide.

SUMMARY:
This study is aim to study the changes of serum creatinine levels at 72 hours after admission in patients with acute heart failure who has diuretic resistance compared to those who do not have diuretic resistance from furosemide stress test

DETAILED DESCRIPTION:
This study is an observational prospective study to demonstrate a prognosis of acute heart failure patients who have diuretic resistance compared to those who do not have diuretic resistance from furosemide stress test. The primary outcome is changes of serum creatinine levels at 72 hours compared to baseline values at the time of admission.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of acute heart failure which is defined by 2 of the 3 following features: ≥2+ leg edema, jugular venous pressure >10 cm from physical examination or central venous pressure >10 mmHg, and bilateral pulmonary edema or bilateral pleural effusion from chest radiography
* Patients consent to participate into the study

Exclusion Criteria:

* Patients who receive furosemide ≥500 mg/day or hydrochlorothiazide ≥100 mg/day or spironolactone ≥100 mg/day or tolvaptan of any doses
* Patients who have systolic blood pressure <100 mmHg or who need vasoactive drugs inotropic agents (except dobutamine)
* Patients with intravascular volume depletion from clinical evaluation
* Patients with chronic kidney disease stage 5 (estimated glomerular filtration rate <15 ml/min/1.73 m2) or patients who receive maintenance dialysis
* Patients who require renal replacement therapy at the time of admission
* Patients whom diagnosed hypertrophic obstructive cardiomyopathy, severe valvular stenosis or complex congenital heart disease
* Patients with sepsis or systemic infection
* Pregnant women
* Patients who have history of furosemide, spironolactone or hydrochlorothiazide allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute heart failure who require intravenous furosemide for the treatment of lung congestion
Sampling Method: Non-Probability Sample
Enrollment: 257 (Estimated)
Dates: Start 2020-07-05 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine | Seventy-two hours after admission
  Changes in serum creatinine from baseline

SECONDARY OUTCOMES:
Serum creatinine | Day 7 of hospital admission
  Changes in serum creatinine from baseline
Requirement for renal replacement therapy | During hospital admission period
  Renal replacement therapy is defined as any mode of dialysis or extracorporeal therapy to treat volume overload for heart failure
Length of hospital admission | During hospital admission period
  Numbers of days that patients need to stay in the hospital
Changes of the stage of heart failure defined by New York Heart Association (NYHA) classification | Day 7 and 28 after hospital admission
  Heart failure stage defined by New York Heart Association (NYHA) classification
Numbers of hospital readmission | Month 1 and 3 after hospital discharge
  Readmission to the hospital due to heart failure
Mortality rate | Day 7 and 28 after hospital admission
  Confirmed death

CONTACTS AND LOCATIONS:
Overall Officials: Kajohnsak Noppakun, MD, Principal Investigator — Instructor, Division of Nephrology, Department of Internal Medicine
Locations (1):
- Chiang Mai University Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Request for individual participant data (IPD) has to be submitted to the Institutional Review Board (IRB) of Faculty of Medicine, Chiang Mai University, Chiang Mai, THAILAND.